CLINICAL TRIAL: NCT00870857
Title: Prevalence and Pathogenesis of Lung Disease in a Large HIV Cohort-coordinating Center
Acronym: MACS
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: University of California, San Francisco (Other); University of Washington (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PRO08050145; 5R01HL090339-02 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-27 (Estimated); Last update posted 2025-08-26 (Actual); Status verified 2016-10

CONDITIONS: HIV Infections; Emphysema; Chronic Obstructive Pulmonary Disease; Pneumocystis
Keywords: Lungs; antiretrovirals; HIV; COPD
MeSH Terms: conditions — HIV Infections; Emphysema; Pulmonary Disease, Chronic Obstructive; Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood oral wash sputum BAL
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Subjects will be 300 HIV+ subjects and 300 HIV- controls selected by random sampling stratified by age and smoking history. Subjects will be recruited from the University of Pittsburgh and the University of Washington (UW) MACS sites. The University of California San Francisco (UCSF) will serve as the recruiting center for the WIHS cohort

SUMMARY:
Despite the availability of highly active antiretroviral therapy (HAART), lung diseases remain a leading cause of morbidity and mortality in those with HIV infection. There have been no large-scale studies detailing pulmonary complications in the HAART era. Substantial gaps exist in our knowledge of the spectrum and pathogenesis of pulmonary disorders in this population, particularly in women and minorities whose numbers with HIV or AIDS have increased. The Multicenter AIDS Cohort Study (MACS) and the Women's Interagency Health Study (WIHS) are prospective, multi-center cohorts that follow approximately 5000 HIV+ subjects and HIV- controls. Although pulmonary disease has not been an area of focus, these established cohorts provide a unique opportunity to systematically study pulmonary complications of HIV infection.

Emphysema is of particular interest in the current HIV era because it is likely to increase as this population lives longer with chronic HIV. HIV-infected persons have an increased incidence of emphysema compared to those without HIV infection, and it has been hypothesized that this accelerated disease progression is the result of one or more latent infectious agents that amplify the pulmonary inflammation. Accelerated emphysema was described in HIV infection in a predominantly male population before HAART. The current prevalence and characteristics of HIV-associated emphysema, and the potential impact of gender, have not been rigorously defined.

DETAILED DESCRIPTION:
HIV-infected patients have an increased incidence of emphysema compared to non-HIV-infected patients, and it has been hypothesized that this accelerated disease progression is the result of one or more latent infections that amplifies the pulmonary inflammatory response. We will examine the prevalence and progression of emphysema in subjects with and without HIV and determine risk factors for emphysema in this population.

Subjects will be 300 HIV+ subjects and 300 HIV- controls selected by random sampling stratified by age and smoking history. Subjects will be recruited from the University of Pittsburgh and the University of California Los Angles (UCLA) MACS sites. The University of California San Francisco (UCSF) will serve as the recruiting center for the WIHS cohort. Because we are interested in an unbiased estimate of the extent of this disease in HIV infection, we will not select subjects based on lung function or current diagnosis of COPD. The HIV- subjects will be matched to the HIV+ subjects in terms of age and smoking history to the extent possible. Those with symptoms of acute respiratory disease such as fevers, acute change in cough or shortness of breath, or weight loss will be excluded. There will be no exclusions based on HAART use or opportunistic infection (OI) prophylaxis and no exclusions based on previous lung disease as we are trying to obtain a comprehensive evaluation of emphysema in this population as well as identify associated risk factors.

All subjects will undergo spirometry, diffusing capacity and quantitative CT scanning. These measurements will allow us to determine differences in the prevalence of emphysema in HIV+ and HIV- and determine risk factors associated with emphysema. For longitudinal studies testing the hypothesis that emphysema is accelerated in HIV infection, we will select HIV+ and HIV- subjects with documented emphysema in each group as defined by diffusing capacity<80% predicted, post-bronchodilator FEV1/FVC<70% without significant reversibility, or at least 10% of lung with a density less than -910 Hounsfield units (HU). These subjects will have CT scans and PFTs at baseline and at 18 months and 36 months after baseline. At each visit, clinical data and biological samples will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Male / Female 18years of age or older.
* Subject has been previously determined to be HIV-infected or is participating in the The Multicenter AIDS Cohort Study (MACS) or the Women's Interagency Health Study (WIHS)

Exclusion Criteria:

* Subject is experiencing acute onset of shortness of breath, cough, fevers or heart conditions problems such as tachycardia, angina or arrhythmias.
* Female subject has told us she is pregnant (this might affect pulmonary function values,we will not require pregnancy testing.)
* Subject has had an MI, CVA, or cardiovascular event within the past 3 months.
* Subject has had eye or abdominal surgery within past 3 months.
* Active TB by documentation or self reported will be exclusion criteria to the study.
* Subjects will be excluded from the study if they are unable to sign consent, weigh > 300 pounds due to technical difficulties with the CT/EBCT scanner, or have been exposed to approximately 10 rads in the previous 12 months (i.e., 2 diagnostic CT scans or 4 cardiac caths or other fluoroscopic exams).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the University of Pittsburgh and the University of California Los Angles MACS sites. The University of California San Francisco will serve as the recruiting center for the WIHS cohort.
Sampling Method: Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2009-01; Primary Completion 2013-10 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
The overall objective of the Pitt coordinating center is to build a collaborative collection of data and specimens that will facilitate the study and understanding of HIV and pulmonary disease | 5 years
  This prospective, multicenter cohort study will survey HIV-infected and non-infected individuals and test for airway obstruction and emphysema and determine associated risk factors. Subjects may be invited back for repeat testing at 18 and 36 months based on the initial test results and measures. Subjects at the multicenter sites may participate in this study for approximately 36 months. Each individual site (University of Pittsburgh, UCLA, UCSF) will be a descriptive longitudinal study to examine the prevalence and progression of emphysema in HIV+ and HIV-subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Morris-Gimbel, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - UCSF, San Francisco, California

REFERENCES:
- [Derived] Cui L, Lucht L, Tipton L, Rogers MB, Fitch A, Kessinger C, Camp D, Kingsley L, Leo N, Greenblatt RM, Fong S, Stone S, Dermand JC, Kleerup EC, Huang L, Morris A, Ghedin E. Topographic diversity of the respiratory tract mycobiome and alteration in HIV and lung disease. Am J Respir Crit Care Med. 2015 Apr 15;191(8):932-42. doi: 10.1164/rccm.201409-1583OC. PMID 25603113